CLINICAL TRIAL: NCT05243563
Title: A Randomized, Unblinded Trial of Topical Steroids Plus CO2 Laser Compared to Steroids Alone in the Treatment of Vulvovaginal Lichen Sclerosus
Brief Title: Does Steroid Plus CO2 Laser Improve Lichen Sclerosus Symptoms Compared to Steroids Alone?
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inability to obtain recruitment levels needed for study to continue.
Sponsor: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1731682-3
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: MonaLisa Touch; fractionated laser; SMARTXIDE2
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Steroids; Clobetasol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractionated CO2 laser plus topical steroids (Experimental): 3 laser treatments at 6 week intervals for 6 months by a single trained operator
  Interventions: Device: MonaLisa Touch; Drug: Topical steroid
- topical steroids alone (Active Comparator): self-applied topical steroid therapy using clobetasol propionate 0.05%
  Interventions: Drug: Topical steroid

INTERVENTIONS:
Device: MonaLisa Touch — 3 laser treatments at 6 week intervals for 6 months by a single trained operator
  Other Names: SMARTXIDE2
  Arms: Fractionated CO2 laser plus topical steroids
Drug: Topical steroid — self-applied topical steroid therapy using clobetasol propionate 0.05%
  Other Names: clobetasol propionate

SUMMARY:
This study will compare the effects of fractionated CO2 laser plus topical steroids versus topical steroids alone in treatment of lichen sclerosus.

DETAILED DESCRIPTION:
Vulvar lichen sclerosus is a common benign skin condition which causes pain and itching. Topical steroids have been the main treatment. A recent study showed that fractionated CO2 laser treatment is non inferior and actually may improve subjective symptoms compared to topical steroids with no serious safety or adverse events. Because steroids reduce risk of vulvar cancer in patients with lichen sclerosus, the investigators hypothesize that steroids in addition to the fractionated laser will provide greater symptom relief while still allowing patient the benefits of steroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with biopsy proven lichen sclerosus and significant symptoms based on Skindex-29 scores >21

Exclusion Criteria:

* prior vaginal mesh or pelvic radiation
* active genital infection
* Current or past gynecologic malignancy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hanes, MD, Principal Investigator — Adjunct Associate Professor of Obstetrics and Gynecology; Stephen Varner, MD, Principal Investigator — Associate Professor of Obstetrics and Gynecology
Locations (2):
- United States (2):
  - USA Health Children's and Women's Hospital, Mobile, Alabama
  - USA Health Strata Patient Center, Mobile, Alabama

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Started | 6 | 5
Completed | 4 | 5
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Skindex-29 Score
Description: The Skindex-29 is a validated tool to assess impact of a chronic skin condition on a person's quality of life. It has been previously used to describe the effects of a treatment and to compare treatments. Values range from 1 (Never) to 5 (All the time). The higher the score, the worse the outcome.
Time Frame: Completed by the subject at baseline and 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 5
Participants
  Decrease in Skindex-29 Score | 3 | 3
  Increase in Skindex-29 Score | 1 | 2

2. Secondary Outcome: Change in Objective Visual Analog Scale
Description: Providers will use this scale to objectively assess vulvar appearance. The tool uses is scored from 0 to 3 (0= absent, 1= mild, 2= moderate, 3= severe) on nine different features of lichen sclerosus (white plaques or hypopigementation, cigarette paper or thin skin, introital narrowing, perianal involvment, loss of labia minora, fusion of labia minora, vulvar fissures, and vulvar erosion). A higher score indicates a higher severity. A higher change in score indicates greater improvement.
Time Frame: Scored by the provider at baseline and 6 months
Population: If scale was not completed at either visit, that participant's data was not included in the outcome measure data.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 4
Participants
  Decrease in score | 3 | 4
  Increase in score | 0 | 0
  No change in score | 1 | 0

3. Secondary Outcome: Change in Vulvovaginal Symptoms Questionnaire (VSQ) Score (Total Score)
Description: This 21 item questionnaire assess four aspects impacting quality of life for patients with vulvovaginal skin diseases: symptoms, emotions, life impact and sexual impact. A higher score corresponds to more bothersome symptoms. The values are 0 (No) or 1 (Yes). The higher the score, the worse the outcome. A higher change in these scores indicates more improvement.
Time Frame: Administered at baseline and at 6 months by the provider.
Population: When scoring the questionnaire, if the participant did not include a score for both the initial and final question, it was not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 5
Participants
  Decrease in score | 4 | 2
  Increase in score | 0 | 2
  No change in score | 0 | 1

4. Secondary Outcome: Change in Vulvovaginal Symptoms Questionnaire Score (Symptoms Component Only)
Description: A subset of the total score on the VSQ, looking at symptoms only. A higher score corresponds to more bothersome symptoms. The values are 0 (No) or 1 (Yes). The higher the score, the worse the outcome. A higher change in these scores indicates more improvement.
Time Frame: Administered at baseline and at 6 months by the provider.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 5
Participants
  Decrease in Score | 3 | 3
  Increase in Score | 1 | 2
  No change in score | 0 | 0

5. Secondary Outcome: Change in Vulvovaginal Symptoms Questionnaire Score (Emotion Component Only)
Description: A subset of the total score on the VSQ, looking at scores for emotions questions only. A higher score corresponds to more emotional impact. The values are 0 (No) or 1 (Yes). The higher the score, the worse the outcome. A higher change in these scores indicates more improvement.
Time Frame: Administered at baseline and at 6 months by the provider.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 5
Participants
  Decrease in score | 3 | 2
  Increase in score | 0 | 3
  No change in score | 1 | 0

6. Secondary Outcome: Change in Vulvovaginal Symptoms Questionnaire Score (Life Impact Component Only)
Description: A subset of the total score on the VSQ, looking at scores for life impact questions only. A higher score corresponds to more impact. The values are 0 (No) or 1 (Yes). The higher the score, the worse the outcome. A higher change in these scores indicates more improvement.
Time Frame: Administered at baseline and at 6 months by the provider.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 5
Participants
  Decrease in score | 2 | 1
  Increase in score | 0 | 1
  No change in score | 2 | 3

7. Secondary Outcome: Change in Vulvovaginal Symptoms Questionnaire Score (Sexual Impact Component Only)
Description: A subset of the total score on the VSQ, looking at scores for sexual impact questions only. A higher score corresponds to more impact. The values are 0 (No) or 1 (Yes). The higher the score, the worse the outcome. A higher change in these scores indicates more improvement.
Time Frame: Administered at baseline and 6 months by an investigator to the subject
Population: Only 1 participant was sexually active at both the initial and final visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 0 | 1
Participants
  No change in score | 0 | 1
  Decrease in score | 0 | 0
  Increase in score | 0 | 0

8. Secondary Outcome: Change in Symptom Subjective Visual Analog Score
Description: This measures the subjects perception of 9 key vulvovaginal symptoms: itching, burning, irritation, pain with intercourse, tearing of vulvar skin, painful urination and painful defecation. Each is scored from 0 -10, with 10 indicating the most symptoms.
Time Frame: Administered at baseline and 6 months by an investigator to the subject
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
Number analyzed (Participants) | 4 | 4
Participants
  Decrease in total score | 3 | 2
  Increase in total score | 1 | 1
  No change in total score | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Reporting Adverse Events Investigators are required to report all AEs experienced by subjects from the time of enrollment until the subject completes the study or terminates early. All AEs, regardless of their relatedness to the study device must be reported. The investigator will evaluate the intensity of the event, severity of the event, and its relatedness to the study device or procedure. All AEs must be followed until resolution or until they become stable.
Arm/Group | Fractionated CO2 Laser Plus Topical Steroids | Topical Steroids Alone
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT05243563/Prot_000.pdf